CLINICAL TRIAL: NCT02170792
Title: Bioavailability of BIBR 953 ZW After Single Oral Doses of 12.5, 50 or 200 mg BIBR 1048 MS Film-coated Tablet Over 2 Days With and Without Coadministration of Ranitidine to Healthy Subjects. Three Groups, 2-way Crossover, Randomised, Open Trial.
Brief Title: Bioavailability of BIBR 953 ZW After Dose of BIBR 1048 MS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1160.16
Record Dates: First submitted 2014-06-20; First posted 2014-06-23 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — Ranitidine

ARMS (2):
- BIBR 1048 MS with ranitidine (Experimental): Low, medium or high dose in combination with ranitidine
  Interventions: Drug: BIBR 1048 MS; Drug: Ranitidine
- BIBR 1048 MS without ranitidine (Experimental): Low, medium or high dose
  Interventions: Drug: BIBR 1048 MS

INTERVENTIONS:
Drug: BIBR 1048 MS — Low, medium or high dose
Drug: Ranitidine — 150mg
  Other Names: Zantic ®
  Arms: BIBR 1048 MS with ranitidine

SUMMARY:
To assess the extent of absorption of 12.5, 50 and 200 mg of BIBR 1048 MS with and without coadministration of 150 mg ranitidine.

ELIGIBILITY:
Inclusion Criteria:

* healthy male subjects as determined by results of screening
* signed written informed consent in accordance with GCP and local legislation
* age >= 18 and <= 50 years
* Broca >= - 20% and <0 + 20%

Exclusion Criteria:

* any finding of the medical examination (including blood pressure, pulse rate and ECG)
* history or current gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic, hormonal disorders
* history of orthostatic hypotension, fainting spells and blackouts
* diseases of central nervous system (such as epilepsy) or psychiatric disorders
* chronic or relevant acute infections
* History of:

  * allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
  * any bleeding disorder including prolonged or habitual bleeding
  * other hematologic disease
  * cerebral bleeding (e.g. after a car accident)
  * commotio cerebri
* intake of drugs with a long half-life (>24 hours) within 1 month prior to administration
* use of any drugs which might influence the results of the trial within 10 days prior to administration or during administration
* participation in another trial with an investigational drug within 2 month prior to administration or during trial
* smoker (> 10 cigarettes or 3 cigars or 3 pipes/day) or inability to refrain from smoking on study days
* alcohol abuse (>60 g / day)
* drug abuse
* blood donation within 1 month prior to administration or during the trial
* excessive physical activities within 5 days prior to administration or during the trial
* any laboratory value outside the clinically accepted reference range
* history of any familial bleeding disorder
* Thrombocytes < 150000 /µl

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2001-02; Primary Completion 2001-03 (Actual)

PRIMARY OUTCOMES:
Area under the plasma drug concentration curve for BIBR 953 ZW from 0 to 12 hours (AUC0-12h) | before and 0.5, 1, 1.5, 2, 4, 6 h after dosing on day 1 and before and 0.5, 1, 1.5, 2, 4, 6, 8, 12 h after dosing on day 2 of each treatment
Area under the plasma drug concentration time curve of BIBR 953 ZW within the interval from zero time to tf (last quantifiable plasma concentration) (AUC0-tf) | before and 0.5, 1, 1.5, 2, 4, 6 h after dosing on day 1 and before and 0.5, 1, 1.5, 2, 4, 6, 8, 12 h after dosing on day 2 of each treatment

SECONDARY OUTCOMES:
Maximum concentration of drug in plasma ( Cmax ) | before and 0.5, 1, 1.5 2, 4, 6 h after dosing on day 1 and before and 0.5, 1, 1.5, 2, 4, 6, 8, 12 h after dosing on day 2 of each treatment
Time from dosing to the maximum concentration of the analyte in plasma (tmax) | before and 0.5, 1, 1.5 2, 4, 6 h after dosing on day 1 and before and 0.5, 1, 1.5, 2, 4, 6, 8, 12 h after dosing on day 2 of each treatment
Changes from baseline in Pulse rate | baseline up to 36 h after last administration
Changes from baseline in blood pressure (systolic and diastolic) | baseline up to 36 h after last administration
Changes from baseline in ECG | baseline up to 36 h after last administration
Changes from baseline in routine laboratory | baseline up to 36 h after last administration
Number of participants with adverse events | up to 36 h after last administration
Changes in international normalized ratio (INR ) | before and 2 hours after treatment
Changes in activated prothrombin time (aPTT) | before and 2 hours after treatment